CLINICAL TRIAL: NCT05259644
Title: The Influence of Laparascopic SLeeve gAstrectomy Vs. Endoscopic Gastric Plication on Body weIght, Metabolic pArameters and Microbiota Composition in Patients With Obesity: Randomized, Open-labelled Study (SLAVIA Trial)
Brief Title: Laparascopic Sleeve Gastrectomy vs. Endoscopic Gastric Plication in Obesity
Acronym: SLAVIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Julius Spicak, prof. MUDr. Julius Spicak, CSc., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NU21-01-00096
Record Dates: First submitted 2022-01-11; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Obesity
Keywords: Obesity; Diabetes mellitus; Endoscopy; Surgery; Gut microbiota
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: In total 75 patients will be randomized into 3 groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative treatment group (Active Comparator): Obese patients treated with conservative approach - diet.
  Interventions: Other: conservative treatment of obesity
- Laparoscopic sleeve gastrectomy (Active Comparator): Obese patients treated with laparoscopic sleeve gastrectomy.
  Interventions: Device: laparoscopic sleeve gastrectomy
- endoscopic gastric plication (Active Comparator): Obese patients treated with endoscopic gastric plication.
  Interventions: Device: endoscopic gastric plication

INTERVENTIONS:
Device: laparoscopic sleeve gastrectomy — Surgical procedure - laparoscopic sleeve gastrectomy.
  Arms: Laparoscopic sleeve gastrectomy
Other: conservative treatment of obesity — Diet and exercise
  Arms: Conservative treatment group
Device: endoscopic gastric plication — Endoscopic procedure - endoscopic gastric plication
  Arms: endoscopic gastric plication

SUMMARY:
The project will describe the efficacy and safety of laparoscopic sleeve gastrectomy and endoscopic gastric plication procedures as compared to conservative therapy and clarify the mechanisms of action of these treatments. The project will also contribute to more precise indications of bariatric or endoscopic methods in clinical practice and enable personalized choice of therapy for particular patient.

DETAILED DESCRIPTION:
Bariatric surgery is the most efficacious treatment of obesity and type 2 diabetes mellitus. Novel endoscopic methods based on the principles of bariatric surgery are also highly effective. No direct randomized comparison of both types of treatment has been performed to date and the mechanisms of action of both procedures are still only partially clarified. The aim of the project is to perform a randomized trial comparing efficacy and safety of three treatment options in patients with obesity: laparoscopic sleeve gastrectomy, endoscopic gastric plication and conservative treatment. A further aim is to characterize the influence of the three treatments on subclinical inflammation, gut microbiota composition and changes of gastrointestinal hormones. The results of the project will describe the efficacy and safety of these procedures as compared to conservative therapy and clarify the mechanisms of action of these treatments. The project will also contribute to more precise indications of bariatric or endoscopic methods in clinical practice and enable personalized choice of therapy for particular patient.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 35 kg/m2
2. For patients with type 2 diabetes - stable antidiabetic medication > 1 month
3. Age 18-60 years

Exclusion Criteria:

1. Other diabetes mellitus types (type 1 DM, monogenic DM, secondary DM)
2. Prior gastrointestinal (GIT) surgery interfering with study procedure
3. Severe gastroesophageal reflux, severe GIT motility disorder
4. Active malignancy
5. Acute myocardial infarction, unstable angina pectoris, acute stroke 3 months prior to enrolment
6. Acute liver or kidney failure
7. Transplantation of insulin producing tissue
8. Gravidity or lactation
9. Mental disorder
10. Inability to sign informed consent
11. Any other contraindication of bariatric surgery or bariatric endoscopy procedure

6. Acute liver or kidney failure 7. Transplantation of insulin producing tissue 8. Gravidity or lactation 9. Mental disorder 10. Inability to sign informed consent 11. Any other contraindication of bariatric surgery or bariatric endoscopy procedure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | 6 months
  To compare the change in body weight after laparoscopic sleeve gastrectomy ve. endoscopic gastric plication and endoscopic gastric plication vs. conservative treatment of obesity

SECONDARY OUTCOMES:
Change in Glycated Hemoglobin | 6 months
  To compare the change in glycated hemoglobin after laparoscopic sleeve gastrectomy ve. endoscopic gastric plication and endoscopic gastric plication vs. conservative treatment of obesity
Change in serum glucagon-like peptide 1 (GLP-1) | 6 months
  To compare the change in serum glucagon-like peptide 1 (GLP-1) after laparoscopic sleeve gastrectomy ve. endoscopic gastric plication and endoscopic gastric plication vs. conservative treatment of obesity
Change in fasting blood glucose | 6 months
  To compare the change in fasting blood glucose after laparoscopic sleeve gastrectomy ve. endoscopic gastric plication and endoscopic gastric plication vs. conservative treatment of obesity

OTHER OUTCOMES:
Change in hsCRP | 6 months
  To compare the change in high sensitive C reactive protein as a marker of low grade inflammation after laparoscopic sleeve gastrectomy and endoscopic gastric plication vs. conservative treatment of obesity
Rehospitalizations | 6 months
  To compare the rate of rehospitalizations after laparoscopic sleeve gastrectomy and endoscopic gastric plication vs. conservative treatment of obesity
Change in the IWQOL (The Impact of Weight on Quality of Life) questionnaire | 6 months
  To compare the change in quality of life as assessed by the IWQOL (The Impact of Weight on Quality of Life) questionnaire after laparoscopic sleeve gastrectomy and endoscopic gastric plication vs. conservative treatment of obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia